CLINICAL TRIAL: NCT00002854
Title: PHASE I PILOT STUDY OF SEQUENTIAL HIGH DOSE CYCLES OF CISPLATIN, CYCLOPHOSPHAMIDE, ETOPOSIDE AND IFOSFAMIDE, CARBOPLATIN AND TAXOL WITH AUTOLOGOUS STEM CELL SUPPORT
Brief Title: High-Dose Combination Chemotherapy Plus Peripheral Stem Cell Transplantation in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 94098; P30CA033572 (NIH); CHNMC-IRB-94098; NCI-V96-1042; CDR0000065102 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Cancer
Keywords: stage IV colon cancer; stage II breast cancer; stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage IV gastric cancer; recurrent gastric cancer; localized osteosarcoma; metastatic osteosarcoma; stage IIIB breast cancer; recurrent pancreatic cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; stage IV anal cancer; recurrent anal cancer; stage IV esophageal cancer; recurrent esophageal cancer; stage III adult soft tissue sarcoma; recurrent adult soft tissue sarcoma; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; recurrent Wilms tumor and other childhood kidney tumors; advanced adult primary liver cancer; recurrent adult primary liver cancer; recurrent osteosarcoma; recurrent gallbladder cancer; recurrent extrahepatic bile duct cancer; recurrent small intestine cancer; stage II melanoma; stage III melanoma; stage IV melanoma; recurrent melanoma; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; stage IV adult soft tissue sarcoma; stage IV pancreatic cancer
MeSH Terms: conditions — Neoplasms; Colonic Neoplasms; Breast Neoplasms; Stomach Neoplasms; Osteosarcoma; Pancreatic Neoplasms; Rectal Neoplasms; Anus Neoplasms; Esophageal Neoplasms; Sarcoma; Carcinoma, Ovarian Epithelial; Wilms Tumor; Carcinoma, Hepatocellular; Gallbladder Neoplasms; Bile Duct Neoplasms; Melanoma; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Filgrastim; Carboplatin; Cisplatin; Cyclophosphamide; Etoposide; Ifosfamide; Mesna; Paclitaxel; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sequential high dose chemotherapy (Experimental)
  Interventions: Biological: filgrastim; Drug: carboplatin; Drug: cisplatin; Drug: cyclophosphamide; Drug: etoposide; Drug: ifosfamide; Drug: mesna; Drug: paclitaxel; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: cisplatin
Drug: cyclophosphamide
Drug: etoposide
Drug: ifosfamide
Drug: mesna
Drug: paclitaxel
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy plus peripheral stem cell transplantation in treating patients who have advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the feasibility of administering 2 courses of high dose chemotherapy consisting of etoposide, cisplatin, and cyclophosphamide followed by ifosfamide, carboplatin, and paclitaxel (IC-T), each administered with filgrastim (G-CSF) and autologous stem cell support, to patients with advanced carcinomas.
* Describe the toxicity of these high dose chemotherapy regimens.
* Define the maximum tolerated dose of paclitaxel deliverable in this high dose regimen.
* Describe the pharmacokinetics of escalating doses of paclitaxel given as a 24-hour continuous infusion.
* Determine the disposition of carboplatin administered in the IC-T regimen.

OUTLINE: At least 4 weeks prior to chemotherapy, patients undergo stem cell collection following filgrastim (G-CSF) mobilization. Sufficient stem cells to support 2 courses of chemotherapy are required. Autologous bone marrow is collected as an adjuvant if stem cell harvest is inadequate.

Patients then receive high dose cisplatin, etoposide, and cyclophosphamide over 10 days, followed the next day by infusion of one fourth of the allotted stem cells, with the remaining allotment infused 2 days later. G-CSF is given for granulocyte support.

Beginning no sooner than 14 weeks from the start of the first course of chemotherapy, stable and responding patients receive high dose paclitaxel, carboplatin, and ifosfamide over 5 days, followed 2 days later with one-fourth of the allotted stem cells, with the remaining allotment infused the following day. G-CSF is given for granulocyte support. Groups of 3-6 patients are treated with escalating doses of paclitaxel until the maximum tolerated dose for this regimen is determined.

Patients are followed monthly for 1 year, every 3 months for 1 year, then as needed at the physician's discretion for at least 5 years.

PROJECTED ACCRUAL: Three to six patients will be entered at each dose of paclitaxel studied.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced carcinomas of the following types:

  * Breast carcinoma that is ineligible for or patient has refused participation in a higher priority protocol in the following categories:

    * Stage II disease with at least 10 involved lymph nodes and no evidence of disease (NED) following surgery
    * Stage III disease rendered surgically NED with or without radiotherapy
    * Stage IV disease following partial response (PR) or complete response (CR) to surgery, chemotherapy, or radiotherapy

      * Prior high dose chemotherapy allowed at discretion of investigator
      * No chemoresistant disease rendered surgically NED
    * Locoregionally recurrent disease within 2 years of breast conservation with or without chemotherapy
* Stage III/IV ovarian cancer

  * PR/CR following debulking surgery and/or chemotherapy
  * Ineligible for or refused participation in higher priority protocols
* Primary soft tissue sarcoma with high-grade disease greater than 10 cm or that is metastatic

  * Rendered surgically NED or achieved PR/CR on any chemotherapeutic or immunotherapeutic regimen
  * Ineligible for or refused participation in higher priority protocols
* Malignant melanoma in the following categories:

  * Ulcerative primary tumor with any number of completely resected metastatic lymph nodes
  * Stage II disease with more than 4 involved nodes rendered NED
  * Stage III disease rendered surgically NED or achieved PR/CR on any chemotherapeutic or immunotherapeutic regimen
* Osteosarcoma that is ineligible for or refused participation in higher priority protocols

  * Resected primary with less than 50% tumor necrosis on pathologic review
  * Metastatic disease rendered surgically NED or PR/CR on any chemotherapeutic, radiotherapeutic, or immunotherapeutic regimen
* The following diseases rendered surgically NED or that achieved PR/CR on any chemotherapeutic, radiotherapeutic, or immunotherapeutic regimen also eligible:

  * Small cell bone carcinoma
  * Metastatic Ewing's sarcoma
  * Metastatic gastrointestinal malignancy
  * Recurrent Wilms' tumor
* No CNS metastases
* No current histologically confirmed bone marrow metastases

  * Prior bone metastases with resolution at time of entry permitted

PATIENT CHARACTERISTICS:

Age:

* Physiologic 18 to 55

Performance status:

* Karnofsky 80%-100%

Hematopoietic:

* Absolute neutrophil count greater than 1,500/mm3
* Platelet count greater than 120,000/mm3
* Hemoglobin greater than 10 g/dL

Hepatic:

* Bilirubin less than 1.5 mg/dL
* AST/ALT less than 3 times normal

Renal:

* Creatinine less than 1.4 mg/dL
* Creatinine clearance at least 70 mL/min
* No history of hemorrhagic cystitis

Cardiovascular:

* Ejection fraction at least 55% by MUGA
* No significant cardiac disease

Pulmonary:

* FEV1 greater than 2 L
* pO2 (room air) greater than 70 mm Hg
* pCO2 (room air) less than 42 mm Hg
* DLCO greater than 60% of predicted

Other:

* No potentially disabling psychosocial history
* No organic or functional CNS dysfunction or other medical problem that would present party at undue risk
* HIV negative
* Hepatitis B surface antigen negative
* No hearing loss greater than 40 decibels
* No contraindication to the following procedures:

  * Collection by apheresis of up to 16 x 10 to the 8th mononuclear cells mobilized by G-CSF
  * Collection of autologous bone marrow, if needed
* No second malignancy except:

  * Nonmelanomatous skin cancer
  * Carcinoma in situ of the cervix
* Not pregnant or nursing
* Adequate contraception required of fertile patients

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* At least 4 weeks since prior immunotherapy

Chemotherapy:

* See Disease Characteristics
* No more than 3 prior chemotherapy regimens (excluding adjuvant therapy)
* No more than 200 mg per square meter of prior cisplatin
* No more than 800 mg per square meter of prior carboplatin
* No prior exposure to greater than 1,000 mg per square meter of "24-hour paclitaxel equivalents" (using a 1:1.3 ratio between paclitaxel doses given by 24-hour infusion and by 3-hour infusion)
* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to more than 20% of bone marrow
* At least 4 weeks since prior radiotherapy

Surgery:

* See Disease Characteristics

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 1994-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Feasibility of two cycles of high dose chemotherapy with stem cell reinfusion | 30 days from start of course II of treatment
Toxicity of two cycles of high dose chemothearpy and stem cell reinfusion | 30 days from start of course II of treatment
  Toxicity graded according to the NCI Common Toxicity Criteria and amended for subjects undergoing transplantation
Maximum tolerated dose of two cycles of high dose chemothearpy and stem cell reinfusion | 30 days from start of course II of treatment

CONTACTS AND LOCATIONS:
Overall Officials: George Somlo, MD, Study Chair — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States